CLINICAL TRIAL: NCT01470092
Title: Double-Blind Randomised Investigation of Tibolone Alone or in Adjunct to Standard Antidepressant Treatment for Depression in Menopausal Women
Brief Title: Tibolone and Placebo in Adjunct to Antidepressant Medication for Women With Menopausal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Professor, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 485/11
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Menopausal Depression
Keywords: Menopause; Depression
MeSH Terms: conditions — Depression | interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tibolone (Active Comparator): Subjects will take 2.5mg of oral Tibolone daily for the duration of the 12 week trial either alone or in adjunct to currently prescribed anti-depressant medication.
  Interventions: Drug: Tibolone
- Placebo (No Intervention): Subjects will take oral placebo tablets packaged daily for the duration of the 12 week trial either alone or in adjunct to currently prescribed antidepressant medication.

INTERVENTIONS:
Drug: Tibolone — Subjects will take 2.5mg of oral Tibolone daily for the duration of the 12 week trial either alone or in adjunct to currently prescribed antidepressant medication.
  Other Names: Livial
  Arms: Tibolone

SUMMARY:
Longitudinal epidemiological studies have shown that many women experience significant physical and psychological changes as they approach menopause and for a long time following. Vasomotor symptoms (such as hot flushes, night sweats), sleep disturbances and changes in libido are common, and impact significantly on the quality of life, social and personal well-being. However, the major reason that many women seek help from menopause clinics or their doctors, is for depression and anxiety symptoms. As such, treatment commonly draws on traditional approaches for the management of major depression including the use of antidepressants such as selective serotonin reuptake inhibitors (SSRIs) or Selective Norepinephrine Reuptake Inhibitors (SNRIs) as the first line response. However, standard treatment of menopausal depression using antidepressants has only shown small improvements at best and at worst, is associated with severe side effects. Some SSRIs have been shown to be less effective in postmenopausal women compared to child bearing age women.

Newer therapies directly targeting the disrupted hormonal systems (in particular estrogen) through the administration of such compounds as tibolone, have shown significant potential to treat depression with the added benefit of fewer adverse side effects. With growing evidence supporting the use of tibolone as a viable and improved treatment for menopausal depression, the investigators propose to investigate the potential of tibolone, a selective Hormone Replacement Therapy (HRT), to ameliorate de-novo or first onset depression occurring in the menopausal period.

DETAILED DESCRIPTION:
All women experience menopause and a significant number suffer from ongoing, severe depression beginning with the major hormone fluctuations in this middle stage of life. Longitudinal epidemiological studies have shown that many women experience significant physical and psychological changes as they approach menopause and for a long time following. Vasomotor symptoms (such as hot flushes, night sweats), sleep disturbances and changes in libido are common, and impact significantly on the quality of life, social and personal well-being. However, the major reason that many women seek help from menopause clinics or their doctors is for depression and anxiety symptoms.

Indeed, many menopausal women with no past psychiatric history experience severe mood symptoms during menopause for the first time in their life, and this has serious and debilitating long term consequences. Treatment for such depression commonly draws on traditional approaches for the management of major depression including the use of antidepressants such as selective serotonin reuptake inhibitors (SSRIs) or selective norepinephrine reuptake inhibitors (SNRIs) as the first line response. However, standard treatment of menopausal depression using antidepressants has only shown small improvements at best and at worst, is associated with severe side effects. Some SSRIs have been shown to be less effective in postmenopausal women compared to women of child bearing age.

Newer therapies directly targeting the fluctuations in reproductive hormonal hormone systems (in particular estrogen, progesterone and testosterone) through the administration of such compounds as tibolone, have shown significant potential to treat depression with the added benefit of fewer adverse side effects. With growing evidence supporting the use of tibolone as a viable and improved treatment for menopausal depression, the investigators propose to investigate the potential of tibolone, a selective Hormone Replacement Therapy (HRT), to ameliorate de-novo or relapsing depression occurring in the menopausal period.

Women with menopausal depression either currently using or not using an SSRI or SNRI medication will be involved in a 12 week randomized control trial in which they may be randomised to one of two groups: i) Tibolone (2.5mg oral/day) or ii) placebo.

It is hypothesized that women receiving Tibolone in adjunct to standard antidepressant medication, will have the same as or a significantly greater improvement in depressive symptoms compared with women receiving placebo in adjunct to standard antidepressant medication and women not using any psychotropic/hormone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females who are currently physically well and between 45 and 65 years of age
* Current DSM-IV diagnosis of depression disorder
* Able to give informed consent
* Menopausal as determined by standardized classification guidelines for female reproductive aging were proposed at the Stages of Reproductive (STRAW) -Aging Workshop and symptom profile on the STRAW
* First-onset or relapse depression during menopause
* Currently taking either an SSRI or SNRI, or no psychotropic medication at all
* Evidence of a normal mammogram in the preceding 12 months.

Exclusion Criteria:

* Patients with known abnormalities in the hypothalamic-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, active or past history of a venous thromboembolic event, breast pathology, undiagnosed vaginal bleeding or abnormal Pap smear results in the previous 2 years.
* Patients with any significant unstable medical illness such as epilepsy and diabetes or known active cardiac, renal or liver disease; or the presence of illness causing immobilisation.
* Patients experiencing severe melancholia, neurovegetative symptoms or current suicidality necessitating acute hospitalisation or intensive psychiatric treatment.
* Patients with psychotic symptoms or past history of severe mental illness including schizophrenia.
* Use of any form of estrogen, progestin or androgen as hormonal therapy, or antiandrogen including Tibolone or use of phytoestrogen supplements as powder or tablet
* Pregnancy / Lactation
* Smoking cigarettes or other nicotine products
* Illicit drug use
* More than 3 standard drinks per day

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale | Baseline, then at weeks 2,4, 8 and 12
  A 10-item clinician rated scale validated to be most strongly sensitive to change in depression associated with treatment. This scale will be used to measure change in depression associated with treatment at weeks 2, 4, 8 and 12 compared to baseline.

SECONDARY OUTCOMES:
The Beck Depression Inventory Second Edition | Baseline and week 12
  A subjective rating scale of depressive symptoms that compliments the MADRS to measure the change of subjective rating of depressive symptoms at week 12 compared to baseline.

OTHER OUTCOMES:
Adverse Symptoms Checklist | Weeks 2, 4, 8 and 12
  A 22 item checklist of general adverse symptoms experienced. This scale will be used to measure adverse symptoms experienced by participants at weeks 2, 4, 8 and 12.
Pittsburgh Sleep Quality Index | Baseline and week 12
  A valid and reliable 19-item self report index measuring sleep quality, latency, duration, disturbances, and daytime dysfunction. This scale will be used to measure different domains of sleep quality at visits occurring at week 12 compared to initial baseline measurement.
Short Form-36 Health Survey (SF-36) | Baseline and week 12
  A 36 item self report measure that assesses: physical health and bodily pain; vitality, social functioning; role limitations due to emotional problems; and mental health. This scale will be used to assess the changes to various domains of self-reported health from baseline compared to week 12.
Menopause Specific Quality of Life Questionnaire | baseline and week 12
  A menopause-specific quality of life questionnaire assessing the presence and severity of vasomotor, psychosocial, physical and sexual symptoms
Menopause Specific Rating Scale for Depression | baseline and week 12
  A 12-item rating scale used to detect depression in menopause.
Hamilton Anxiety Scale | Baseline and weeks 2,4,8 and 12
  A 14-item scale used to assess the severity of anxiety symptoms.
Sexual Interest and Desire Inventory | Baseline and week 12
  A 13 item measure of the severity of symptoms related to hypoactive sexual desire

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, PhD,FRANZP, Principal Investigator — Monash Alfred Psychiatry Research Centre
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulkarni J, Gavrilidis E, Thomas N, Hudaib AR, Worsley R, Thew C, Bleeker C, Gurvich C. Tibolone improves depression in women through the menopause transition: A double-blind randomized controlled trial of adjunctive tibolone. J Affect Disord. 2018 Aug 15;236:88-92. doi: 10.1016/j.jad.2018.04.103. Epub 2018 Apr 24. PMID 29723767